CLINICAL TRIAL: NCT03854279
Title: Bizact Versus Electroscissor for Adult Tonsillectomy
Brief Title: Comparison of Bizact With Electroscissor for Tonsillectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Johan C Ræder, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bizact study
Record Dates: First submitted 2019-02-23; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Tonsillar Hypertrophy, Tonsillitis
MeSH Terms: conditions — Tonsillitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bizact (Experimental): Tonsillectomy will be done With the Bizact device
  Interventions: Device: tonsillar dissection
- Electro-scissor (Active Comparator): Tonsillectomy will be done With electro-scissors
  Interventions: Device: tonsillar dissection

INTERVENTIONS:
Device: tonsillar dissection — The tonsils will be removed by bizact device

SUMMARY:
In a randomized, partly double-blind prospective setup we want to compare traditional adult electro-scissor tonsillectomy With ultrasound Technology, Bizact.

ELIGIBILITY:
Inclusion Criteria:

* planned elective tonsillectomy
* informed consent

Exclusion Criteria:

* regular use of analgesics pre-operatively
* known tendency of bleeding
* not able to communicate in Norwegian

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain: Number of days With need of analgesics | 2 weeks
  Number of days With need of analgesics

SECONDARY OUTCOMES:
Postoperative pain: Dose need of pain killers during first 24 hr postoperatively | 24 hrs
  Dose need of pain killers during first 24 hr postoperatively
Postoperative bleeding | 2 weeks
  Incidence of bleeding after discharge
Per-operative bleeding | per-operative
  Amount of bleeding during surgery
Duration of surgery | 0 - 1 hr
  time from start of surgery to end

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Anesthesiology, Oslo University Hospital, Ullevaal, Oslo, Norway